CLINICAL TRIAL: NCT00415701
Title: Effect of an Anesthetic Induction Dose of Etomidate on Hemodynamics and Adrenocortical Function After Cardiac Surgery
Brief Title: Effect of Etomidate on Hemodynamics and Adrenocortical Function After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Stefan M Jakob, Professor, Department of Critical Care Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DINA-KEK7406-IBAN-2006-1
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Disease; Mitral Valve Regurgitation
Keywords: Etomidate; Propofol; Adrenocortical Insufficiency; Hemodynamic Process; Vasoactive Agonists; Coronary Artery Bypass; Ischemic Coronary Heart Disease; Mitral valve reconstruction/replacement; Mitral valve regurgitation; Heart Valve Prosthesis; Cardiopulmonary Bypass
MeSH Terms: conditions — Coronary Artery Disease; Mitral Valve Insufficiency; Addison Disease | interventions — Etomidate; Propofol; Hydrocortisone; Sodium Chloride; Cosyntropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Etomidate as a single induction dose
  Interventions: Drug: Etomidate
- 2 (Active Comparator): Propofol as a single induction dose
  Interventions: Drug: Propofol
- 3 (Other): Hydrocortisone substitution or placebo (50-50%) in etomidate-group
  Interventions: Drug: Hydrocortisone; Drug: NaCl 0.9%; Other: Tetracosactin

INTERVENTIONS:
Drug: Etomidate — Single induction dose of etomidate 0.2%; total dose 0.15 mg/kg
  Arms: 1
Drug: Propofol — Single induction dose of propofol 2%; total dose 1.5 mg/kg
  Arms: 2
Drug: Hydrocortisone — Hydrocortisone 100 mg/2 ml: day of operation 3x, POD 1 2x, POD 2 1x
  Arms: 3
Drug: NaCl 0.9% — NaCl 0.9% 2 ml; day of operation 3x, POD 1 2x, POD 2 1x
  Arms: 3
Other: Tetracosactin — Diagnostic test, Tetracosactin 250 microg iv
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effect of a single dose of etomidate for patients undergoing cardiac surgery with the use of cardiopulmonary bypass (CPB) on post-CPB adrenocortical responsiveness, on requirements of hemodynamic support, and on use of intensive care resources.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients undergoing elective

  * coronary artery bypass graft (primary or re-operation)
  * mitral valve reconstruction/replacement for mitral valve regurgitation
* Age between 18 and 80 years (extremes included)
* Subject itself has signed the informed consent
* No clinically relevant deviation from the laboratory's reference range of biochemistry, hematology, or urinalysis testing

Exclusion Criteria:

* Participation in another ongoing interventional trial
* Known adrenocortical insufficiency
* Use of etomidate or propofol within 1 week preoperatively
* Use of glucocorticoids within 6 month preoperatively
* Known sensitivity to etomidate, propofol, or emulgator
* Severe hepatic dysfunction (bilirubin > 3mg/dl)
* Severe renal dysfunction (plasma creatinine > 180mikromol/l)
* Sepsis, endocarditis or other chronic inflammatory disease
* Manifest insulin-dependent diabetes mellitus
* Positive HIV serology
* Hemodynamically significant carotid stenosis requiring treatment
* Serious illnesses: endocrine, neurological, psychiatric, metabolic disturbances
* Pregnancy or breast-feeding female; females will be subject to pregnancy testing
* Requirement of rapid sequence induction
* Emergency surgery
* History of asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of absolute and relative adrenal insufficiency | Preoperative day to postoperative day (POD) 4
Cumulative requirements of vasoactive drugs during surgery and in the intensive care unit (ICU) | Induction of anesthesia to POD 2

SECONDARY OUTCOMES:
Incidence of failure to wean off cardiopulmonary bypass on first intention | intraoperatively
Serum lactate | Induction of anesthesia to discharge ICU
Time to extubation | Induction of anesthesia to extubation
Length of stay (LOS) in the intensive care unit (ICU), intermediate care unit (IMC), and hospital | Admission to discharge: ICU, IMC, and hospital
Association of results with preoperative risk, stress-dose hydrocortisone replacement, type of surgery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Jakob, Professor, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Departments of Intensive Care Medicine and Anesthesiology, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Malerba G, Romano-Girard F, Cravoisy A, Dousset B, Nace L, Levy B, Bollaert PE. Risk factors of relative adrenocortical deficiency in intensive care patients needing mechanical ventilation. Intensive Care Med. 2005 Mar;31(3):388-92. doi: 10.1007/s00134-004-2550-8. Epub 2005 Feb 10. PMID 15703896
- [Background] Weis F, Kilger E, Roozendaal B, de Quervain DJ, Lamm P, Schmidt M, Schmolz M, Briegel J, Schelling G. Stress doses of hydrocortisone reduce chronic stress symptoms and improve health-related quality of life in high-risk patients after cardiac surgery: a randomized study. J Thorac Cardiovasc Surg. 2006 Feb;131(2):277-82. doi: 10.1016/j.jtcvs.2005.07.063. PMID 16434254
- [Background] den Brinker M, Joosten KF, Liem O, de Jong FH, Hop WC, Hazelzet JA, van Dijk M, Hokken-Koelega AC. Adrenal insufficiency in meningococcal sepsis: bioavailable cortisol levels and impact of interleukin-6 levels and intubation with etomidate on adrenal function and mortality. J Clin Endocrinol Metab. 2005 Sep;90(9):5110-7. doi: 10.1210/jc.2005-1107. Epub 2005 Jun 28. PMID 15985474
- [Background] Absalom A, Pledger D, Kong A. Adrenocortical function in critically ill patients 24 h after a single dose of etomidate. Anaesthesia. 1999 Sep;54(9):861-7. doi: 10.1046/j.1365-2044.1999.01003.x. PMID 10460557
- [Background] Annane D. ICU physicians should abandon the use of etomidate! Intensive Care Med. 2005 Mar;31(3):325-6. doi: 10.1007/s00134-005-2560-1. Epub 2005 Jan 27. No abstract available. PMID 15750800
- [Background] Duthie DJ, Fraser R, Nimmo WS. Effect of induction of anaesthesia with etomidate on corticosteroid synthesis in man. Br J Anaesth. 1985 Feb;57(2):156-9. doi: 10.1093/bja/57.2.156. PMID 2982387
- [Background] Fellows IW, Bastow MD, Byrne AJ, Allison SP. Adrenocortical suppression in multiply injured patients: a complication of etomidate treatment. Br Med J (Clin Res Ed). 1983 Dec 17;287(6408):1835-7. doi: 10.1136/bmj.287.6408.1835. PMID 6322902
- [Background] Fellows IW, Byrne AJ, Allison SP. Adrenocortical suppression with etomidate. Lancet. 1983 Jul 2;2(8340):54-5. doi: 10.1016/s0140-6736(83)90043-0. No abstract available. PMID 6134923
- [Background] Wagner RL, White PF, Kan PB, Rosenthal MH, Feldman D. Inhibition of adrenal steroidogenesis by the anesthetic etomidate. N Engl J Med. 1984 May 31;310(22):1415-21. doi: 10.1056/NEJM198405313102202. PMID 6325910
- [Background] Allolio B, Stuttmann R, Fischer H, Leonhard W, Winkelmann W. Long-term etomidate and adrenocortical suppression. Lancet. 1983 Sep 10;2(8350):626. doi: 10.1016/s0140-6736(83)90710-9. No abstract available. PMID 6136774
- [Background] Crozier TA, Beck D, Wuttke W, Kettler D. [Relation of the inhibition of cortisol synthesis in vivo to plasma etomidate concentrations]. Anaesthesist. 1988 May;37(5):337-9. German. PMID 3261141
- [Background] Watt I, Ledingham IM. Mortality amongst multiple trauma patients admitted to an intensive therapy unit. Anaesthesia. 1984 Oct;39(10):973-81. doi: 10.1111/j.1365-2044.1984.tb08885.x. PMID 6496912
- [Background] Kenyon CJ, McNeil LM, Fraser R. Comparison of the effects of etomidate, thiopentone and propofol on cortisol synthesis. Br J Anaesth. 1985 May;57(5):509-11. doi: 10.1093/bja/57.5.509. PMID 2986663
- [Background] Kilger E, Weis F, Briegel J, Frey L, Goetz AE, Reuter D, Nagy A, Schuetz A, Lamm P, Knoll A, Peter K. Stress doses of hydrocortisone reduce severe systemic inflammatory response syndrome and improve early outcome in a risk group of patients after cardiac surgery. Crit Care Med. 2003 Apr;31(4):1068-74. doi: 10.1097/01.CCM.0000059646.89546.98. PMID 12682474
- [Background] Loisa P, Uusaro A, Ruokonen E. A single adrenocorticotropic hormone stimulation test does not reveal adrenal insufficiency in septic shock. Anesth Analg. 2005 Dec;101(6):1792-1798. doi: 10.1213/01.ANE.0000184042.91452.48. PMID 16301260
- [Background] Neumann R, Worek FS, Blumel G, Zimmermann GJ, Fehm HL, Pfeiffer UJ. Cortisol deficiency in metomidate anesthetized bacteremic pigs: results in circulatory failure--beneficial effect of cortisol substitution. Acta Anaesthesiol Scand. 1989 Jul;33(5):379-84. doi: 10.1111/j.1399-6576.1989.tb02927.x. PMID 2572134
- [Derived] Basciani RM, Rindlisbacher A, Begert E, Brander L, Jakob SM, Etter R, Carrel T, Eberle B. Anaesthetic induction with etomidate in cardiac surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jun;33(6):417-24. doi: 10.1097/EJA.0000000000000434. PMID 26914224